CLINICAL TRIAL: NCT01349816
Title: A Randomized, Double Blind, Chronic Dosing (7 Days), Two Period, Six Treatment, Incomplete Block, Cross Over, Multi Center Study to Assess Efficacy and Safety of Four Doses of PT003 MDI in Patients With Moderate to Severe COPD, Compared With Its Individual Components (PT005 MDI and PT001 MDI) as Active Controls
Brief Title: PT003 MDI Dose Confirmation Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pearl Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PT003004
Record Dates: First submitted 2011-05-05; First posted 2011-05-09 (Estimated); Results first posted 2017-04-27 (Actual); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- PT003 (Dose 1) (Experimental): PT003 MDI Dose 1
  Interventions: Drug: PT003
- PT003 (Dose 2) (Experimental): PT003 MDI Dose 2
  Interventions: Drug: PT003
- PT003 (Dose 3) (Experimental): PT003 MDI Dose 3
  Interventions: Drug: PT003
- PT003 (Dose 4) (Experimental): PT003 MDI Dose 4
  Interventions: Drug: PT003
- PT001 (Experimental): PT001 MDI
  Interventions: Drug: PT001
- PT005 (Experimental): PT005 MDI
  Interventions: Drug: PT005

INTERVENTIONS:
Drug: PT003 — PT003 MDI administered as two puffs BID for 7 days
  Arms: PT003 (Dose 1); PT003 (Dose 2); PT003 (Dose 3); PT003 (Dose 4)
Drug: PT001 — PT001 MDI administered as two puffs BID for 7 days
  Arms: PT001
Drug: PT005 — PT005 MDI administered as two puffs BID for 7 days
  Arms: PT005

SUMMARY:
The primary objective of this study is to demonstrate efficacy of PT003 MDI relative to its individual components (PT001 MDI and PT005 MDI) in patients with moderate to severe chronic obstructive pulmonary disease (COPD).

ELIGIBILITY:
Key Inclusion Criteria:

* Signed written informed consent
* 40 - 80 years of age
* Clinical history of COPD with airflow limitation that is not fully reversible
* Females of non-child bearing potential or females of child bearing potential with negative pregnancy test; and acceptable contraceptive methods
* Current/former smokers with at least a 10 pack-year history of cigarette smoking
* A measured post- bronchodilator FEV1/FVC ratio of < or = 0.70
* A measured post- bronchodilator FEV1 > or = 750ml or 30% predicted and < or = 80% of predicted normal values
* Able to change COPD treatment as required by protocol

Key Exclusion Criteria:

* Women who are pregnant or lactating
* Primary diagnosis of asthma
* Alpha-1 antitrypsin deficiency as the cause of COPD
* Active pulmonary diseases
* Prior lung volume reduction surgery
* Abnormal chest X-ray (or CT scan) not due to the presence of COPD
* Hospitalized due to poorly controlled COPD within 3 months of Screening
* Clinically significant medical conditions that preclude participation in the study (e.g. clinically significant abnormal ECG, uncontrolled hypertension, glaucoma, symptomatic prostatic hypertrophy)
* Cancer that has not been in complete remission for at least 5 years
* Treatment with investigational study drug or participation in another clinical trial or study within the last 30 days or 5 half lives

Other inclusion/exclusion criteria as defined in the protocol

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2011-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colin Reisner, M.D., Study Director — Pearl Therapeutics, Inc.
Locations (13):
- United States (13):
  - Pearl Investigative Site, Rancho Mirage, California
  - Pearl Investigative Site, Colorado Springs, Colorado
  - Pearl Investigative Site, Waterbury, Connecticut
  - Pearl Investigative Site, Clearwater, Florida
  - Pearl Investigative Site, Pensacola, Florida
  - Pearl Investigative Site, Stockbridge, Georgia
  - Pearl Investigative Site, Minneapolis, Minnesota
  - Pearl Investigative Site, Brooklyn, New York
  - Pearl Investigative Site, Charlotte, North Carolina
  - Pearl Investigative Site, Winston-Salem, North Carolina
  - Pearl Investigative Site, Cincinnati, Ohio
  - Pearl Investigative Site, Medford, Oregon
  - Pearl Investigative Site, Spartanburg, South Carolina

REFERENCES:
- [Derived] Reisner C, Pearle J, Kerwin EM, Rose ES, Darken P. Efficacy and safety of four doses of glycopyrrolate/formoterol fumarate delivered via a metered dose inhaler compared with the monocomponents in patients with moderate-to-severe COPD. Int J Chron Obstruct Pulmon Dis. 2018 Jun 19;13:1965-1977. doi: 10.2147/COPD.S166455. eCollection 2018. PMID 29950826

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Conducted at 14 US sites from July-November 2011. Entire study period of study participation was a maximum of 9 weeks.
Pre-assignment Details: Study was a chronic dosing study; each participant received 2 of 6 possible treatments; each treatment period was separated by a washout period of at least 7 days. Patients were randomized into one of 30 treatment sequences. Each sequence included exactly 2 of the 6 treatment groups for this study.
Groups:
- Overall Study: Overall Study
Period: Overall Study
Arm/Group | Overall Study
Started | 185
GP MDI 36 µg | 61
GFF MDI 36/7.2 µg | 58
GFF MDI 36/9.6 µg | 56
GFF MDI 18/9.6 µg | 57
GFF MDI 9/9.6 µg | 57
FF MDI 9.6 µg | 61
Completed | 155
Not Completed | 30
Not completed — Withdrawal by Subject | 4
Not completed — Physician Decision | 1
Not completed — Adverse Event | 14
Not completed — Lost to Follow-up | 2
Not completed — Protocol Violation | 1
Not completed — Protocol-specified criteria | 8

BASELINE CHARACTERISTICS:
Population: Analysis population included all randomized subjects
Groups:
- Overall Study: All patients randomized and treated
Arm/Group | Overall Study
Number analyzed (Participants) | 185
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.1 (9.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78
  Male | 107

OUTCOME MEASURES:

1. Primary Outcome: FEV1 AUC0-12
Description: Forced Expiratory Volume in One Second (FEV1) Area Under the Curve (AUC) 0-12 relative to baseline following chronic dosing (1 week).
Time Frame: Day 7
Population: Modified Intent to Treat (MITT) Population is made of participants who completed both treatment periods and had Pre-dose Day 1 data for both and no protocol deviations believed to have a potential impact on efficacy results. Subjects must have had data for the given endpoint to be included.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Groups:
- GFF MDI 36/7.2 µg: GFF MDI 36/7.2 µg BID
- GFF MDI 36/9.6 µg: GFF MDI 36/9.6 µg BID
- GFF MDI 18/9.6 µg: GFF MDI 18/9.6 µg BID
- GFF MDI 9/9.6 µg: GFF MDI 9/9.6 µg BID
- GP MDI 36 µg: GP MDI 36 µg BID
- FF MDI 9.6 µg: FF MDI 9.6 µg BID
Arm/Group | GFF MDI 36/7.2 µg | GFF MDI 36/9.6 µg | GFF MDI 18/9.6 µg | GFF MDI 9/9.6 µg | GP MDI 36 µg | FF MDI 9.6 µg
Number analyzed (Participants) | 49 | 42 | 44 | 50 | 49 | 50
Liters | 1.467 [1.424 to 1.511] | 1.462 [1.418 to 1.508] | 1.493 [1.448 to 1.539] | 1.499 [1.455 to 1.544] | 1.399 [1.358 to 1.441] | 1.465 [1.423 to 1.509]

2. Secondary Outcome: Peak Change From Baseline in FEV1
Description: Peak change from baseline in FEV1 through 2 hours
Time Frame: Day 1
Population: MITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | GFF MDI 36/7.2 µg | GFF MDI 36/9.6 µg | GFF MDI 18/9.6 µg | GFF MDI 9/9.6 µg | GP MDI 36 µg | FF MDI 9.6 µg
Number analyzed (Participants) | 49 | 43 | 45 | 52 | 51 | 51
Liters | 0.312 [0.265 to 0.359] | 0.308 [0.259 to 0.358] | 0.344 [0.295 to 0.393] | 0.350 [0.304 to 0.397] | 0.248 [0.201 to 0.294] | 0.307 [0.260 to 0.353]

3. Secondary Outcome: Time to Onset of Action
Description: At least 10% improvement in mean FEV1
Time Frame: Day 1
Population: MITT Population
Measure: Number; unit: Participants
Arm/Group | GFF MDI 36/7.2 µg | GFF MDI 36/9.6 µg | GFF MDI 18/9.6 µg | GFF MDI 9/9.6 µg | GP MDI 36 µg | FF MDI 9.6 µg
Number analyzed (Participants) | 50 | 43 | 45 | 52 | 51 | 51
Participants
  15 minutes | 28 [0.265 to 0.359] | 21 [0.259 to 0.358] | 20 [0.295 to 0.393] | 30 [0.304 to 0.397] | 15 [0.201 to 0.294] | 24 [0.260 to 0.353]
  30 minutes | 10 | 9 | 8 | 8 | 14 | 14
  1 hour | 4 | 3 | 9 | 5 | 7 | 6
  2 hours | 4 | 2 | 2 | 3 | 3 | 2
  No onset within 2 hours | 4 | 8 | 6 | 6 | 12 | 5

4. Secondary Outcome: At Least 12% Improvement in FEV1
Description: Proportion of subjects achieving >=12% improvement in FEV1 relative to baseline
Time Frame: Day 1
Population: MITT Population
Measure: Number; unit: Participants
Arm/Group | GFF MDI 36/7.2 µg | GFF MDI 36/9.6 µg | GFF MDI 18/9.6 µg | GFF MDI 9/9.6 µg | GP MDI 36 µg | FF MDI 9.6 µg
Number analyzed (Participants) | 50 | 43 | 45 | 52 | 51 | 51
Participants
  15 minutes | 22 [0.265 to 0.359] | 17 [0.259 to 0.358] | 18 [0.295 to 0.393] | 27 [0.304 to 0.397] | 13 [0.201 to 0.294] | 22 [0.260 to 0.353]
  30 minutes | 14 | 10 | 8 | 7 | 12 | 10
  1 hour | 2 | 5 | 6 | 4 | 5 | 7
  2 hours | 2 | 3 | 5 | 6 | 4 | 5
  No onset within 2 hours | 10 | 8 | 8 | 8 | 17 | 7

5. Secondary Outcome: Peak Change in IC
Description: Mean inspiratory capacity (IC) of 1 and 2 hours post-dose minus baseline
Time Frame: Day 1
Population: MITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | GFF MDI 36/7.2 µg | GFF MDI 36/9.6 µg | GFF MDI 18/9.6 µg | GFF MDI 9/9.6 µg | GP MDI 36 µg | FF MDI 9.6 µg
Number analyzed (Participants) | 48 | 43 | 45 | 52 | 51 | 51
Liters | 0.323 [0.249 to 0.397] | 0.242 [0.165 to 0.319] | 0.339 [0.264 to 0.415] | 0.326 [0.254 to 0.398] | 0.228 [0.156 to 0.300] | 0.316 [0.244 to 0.388]

6. Secondary Outcome: Morning Pre-dose FEV1
Description: Change from baseline in morning pre-dose FEV1 (average of 60- and 30-minute pre-dose values on Day 7)
Time Frame: Day 7
Population: MITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | GFF MDI 36/7.2 µg | GFF MDI 36/9.6 µg | GFF MDI 18/9.6 µg | GFF MDI 9/9.6 µg | GP MDI 36 µg | FF MDI 9.6 µg
Number analyzed (Participants) | 49 | 43 | 45 | 52 | 51 | 51
Liters | 0.152 [0.105 to 0.199] | 0.110 [0.061 to 0.159] | 0.122 [0.073 to 0.170] | 0.131 [0.085 to 0.177] | 0.100 [0.053 to 0.146] | 0.103 [0.057 to 0.149]

7. Secondary Outcome: FEV1 Through 6 Hours
Description: Peak change from baseline in FEV1 through 6 hours
Time Frame: Day 7
Population: MITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | GFF MDI 36/7.2 µg | GFF MDI 36/9.6 µg | GFF MDI 18/9.6 µg | GFF MDI 9/9.6 µg | GP MDI 36 µg | FF MDI 9.6 µg
Number analyzed (Participants) | 50 | 42 | 45 | 51 | 51 | 51
Liters | 0.362 [0.309 to 0.414] | 0.356 [0.300 to 0.412] | 0.388 [0.334 to 0.443] | 0.415 [0.363 to 0.467] | 0.283 [0.231 to 0.336] | 0.355 [0.302 to 0.408]

8. Secondary Outcome: Peak Change From Baseline in IC
Description: Peak change from baseline in inspiratory capacity (IC) (mean of 1 and 2 hours post-dose minus baseline)
Time Frame: Day 7
Population: MITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | GFF MDI 36/7.2 µg | GFF MDI 36/9.6 µg | GFF MDI 18/9.6 µg | GFF MDI 9/9.6 µg | GP MDI 36 µg | FF MDI 9.6 µg
Number analyzed (Participants) | 48 | 43 | 45 | 52 | 51 | 51
Liters | 0.333 [0.246 to 0.420] | 0.267 [0.177 to 0.357] | 0.340 [0.252 to 0.429] | 0.351 [0.267 to 0.436] | 0.228 [0.143 to 0.313] | 0.354 [0.269 to 0.439]

9. Secondary Outcome: Mean Evening Trough FEV1
Description: Change from baseline in mean evening 12-hour post-dose trough FEV1
Time Frame: Day 7
Population: MITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | GFF MDI 36/7.2 µg | GFF MDI 36/9.6 µg | GFF MDI 18/9.6 µg | GFF MDI 9/9.6 µg | GP MDI 36 µg | FF MDI 9.6 µg
Number analyzed (Participants) | 48 | 43 | 44 | 51 | 49 | 50
Liters | 0.080 [0.032 to 0.129] | 0.073 [0.023 to 0.123] | 0.105 [0.055 to 0.154] | 0.112 [0.064 to 0.159] | 0.081 [0.033 to 0.129] | 0.120 [0.073 to 0.168]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the subject signed consent up to the follow-up (Final) visit or premature discontinuation visit.
Description: Safety population included all participants who received at least one dose of study drug, with safety data available. Serious adverse events were collected from the time the subject signed consent up to 14 days following the last dose of study drug.
Arm/Group | GFF MDI 36/7.2 µg | GFF MDI 36/9.6 µg | GFF MDI 18/9.6 µg | GFF MDI 9/9.6 µg | GP MDI 36 µg | FF MDI 9.6 µg
Serious Adverse Events (participants affected / at risk) | 1/58 | 0/56 | 0/57 | 0/57 | 2/61 | 0/61
Other Adverse Events (participants affected / at risk) | 9/58 | 4/56 | 1/57 | 7/57 | 2/61 | 8/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GFF MDI 36/7.2 µg (N=58) | GFF MDI 36/9.6 µg (N=56) | GFF MDI 18/9.6 µg (N=57) | GFF MDI 9/9.6 µg (N=57) | GP MDI 36 µg (N=61) | FF MDI 9.6 µg (N=61)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GFF MDI 36/7.2 µg (N=58) | GFF MDI 36/9.6 µg (N=56) | GFF MDI 18/9.6 µg (N=57) | GFF MDI 9/9.6 µg (N=57) | GP MDI 36 µg (N=61) | FF MDI 9.6 µg (N=61)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 3 (3) | 1 (1) | 5 (5) | 2 (2) | 4 (4)
Tremor (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (4)
Headache (Nervous system disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Drafts of any and all publications or presentations of this study must be submitted at least 30 days prior to submission for publication or presentation to Pearl Therapeutics for review, approval, and to ensure consistency. Pearl Therapeutics has the right to request appropriate modification to correct facts and to represent its opinions, or the opinions of the publication committee, if these differ with the proposed publication.